CLINICAL TRIAL: NCT01449214
Title: Ultrasound-Guided Technique for Thoracic Epidural Insertion: A Randomized Controlled Trial
Brief Title: Ultrasound-Guided Technique for Thoracic Epidural Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-03
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Pain
Keywords: Thoracic epidural; Epidural anesthesia; Ultrasound; Palpation; Thoracic spine
MeSH Terms: conditions — Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): Use of ultrasound to identify interlaminar spaces for needle insertion. Intervention/Procedure: ultrasound-guided technique.
  Interventions: Procedure: Ultrasound
- Landmarking (Active Comparator): Use of manual palpation to identify anatomic landmarks for needle insertion. Procedure/Intervention: landmark-guided technique.
  Interventions: Procedure: Landmarking

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound-guided technique
  Arms: Ultrasound
Procedure: Landmarking — Landmark-guided technique
  Arms: Landmarking

SUMMARY:
Thoracic epidural analgesia and anesthesia are effective in improving the quality of intraoperative and postoperative pain relief during thoracic and abdominal surgical procedures. Conventional epidural techniques have significant limitations. Due to the anatomic characteristics of the thoracic versus the lumbar intervertebral spaces, the insertion requires a more technically challenging paramedian approach. The safety and feasibility of bedside ultrasonography for the lumbar spine has already been established and it proves to be a valuable tool for neuraxial anesthesia in obstetric anesthesia

DETAILED DESCRIPTION:
• The feasibility and the reliability of US imaging for the thoracic spine has been proven by comparing the findings of ultrasound scans to MRI measurements, which is the standard imaging technique for the depiction of the spine. Pre-puncture US assessment may contribute to the safety and efficacy of the thoracic epidural technique. The purpose of this study is to compare the ultrasound-guided thoracic epidural insertion technique with the conventional anatomic landmarking technique of contacting bone and walking-off the lamina

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Elective major abdominal or thoracic surgery requiring thoracic epidural anesthesia/analgesia.
* Consent to participate and signed consent form.

Exclusion Criteria:

* Contraindication to epidural anesthesia.
* Marked spinal deformities or a history of spinal instrumentation
* Emergency surgery.
* Inability to communicate in English.
* BMI>35 kgm-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Needle redirections | 30 minutes
  Number of needle redirections defined as the need to withdraw the epidural needle for the purpose of continuing on a different angle (sagittal or axial plane)

SECONDARY OUTCOMES:
Bony contacts | 30 minutes
  number of bony contacts during the needle insertion
New insertion point | 30 minutes
  need to re-insert the epidural needle in the same interlaminar space, but using different insertion point
Number of insertions | 30 minutes
  number of different interlaminar space insertions
duration of ultrasound scanning | 30 minutes
  duration of ultrasound scanning
duration of epidural procedure | 30 minutes
  duration of epidural procedure
complications during epidural insertion | 30 minutes
  complications during epidural insertion

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Arzola, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (2):
- Canada (2):
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario